CLINICAL TRIAL: NCT02623127
Title: A Phase II, Non-comparative, Open Label, Multi-center Study of Sunitinib in Patients With Metastatic or Recurrent Thymic Carcinoma
Brief Title: A Study of Sunitinib in Patients With Metastatic or Recurrent Thymic Carcinoma
Acronym: KOSMIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Seok Lee, Professor of Internal Medicine, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-15-01
Record Dates: First submitted 2015-10-28; First posted 2015-12-07 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Thymic Carcinoma
Keywords: Thymic carcinoma; Sunitinib; Metastatic; Recurrent
MeSH Terms: conditions — Thymoma; Neoplasm Metastasis; Recurrence | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib (Experimental): Sunitinib will be administered orally at a dose of 50 mg once daily in 3-week cycles consisting of 2 weeks of treatment followed by 1 week without treatment.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib

SUMMARY:
This study aims to investigate the clinical activity of sunitinib in patients with advanced thymic carcinoma who have failed chemotherapy.

DETAILED DESCRIPTION:
Sunitinib (Sutent®; Pfizer, New York, NY, USA) is a multitargeted tyrosine-kinase inhibitor (TKI) with activity against the stem cell-factor receptor (KIT) and platelet-derived growth-factor receptor (PDGFR), vascular endothelial growth-factor receptor (VEGFR), glial cell line-derived neurotrophic factor receptor (rearranged during transfection [RET]), colony-stimulating factor-1 receptor (CSF1R), and Fms-like tyrosine kinase-3 receptor (FLT3).

Sunitinib is a potent inhibitor of mutant KIT with additional inhibitory effects on VEGF receptors that potentially might make it more effective than imatinib against TCs. In the current version of NCCN guideline, sunitinib is suggested as one of the potential targeted therapeutics for advanced TCs.

We planned this study to investigate the clinical efficacy and tolerability of sunitinib in patients with advanced or recurrent TCs in Korean population. In addition, we will collect tumor samples and blood samples from patients for the further exploration of predictive biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed, written and dated informed consent prior to any study specific procedures
2. Histopathologically confirmed metastatic or recurrent thymic thymic carcinoma
3. Age ≥ 20
4. ECOG PS 0-2
5. Documented progressive disease after one or more conventional systemic chemotherapy
6. At least one measurable disease by RECIST v1.1
7. Adequate organ function for treatment as follows:

   * Absolute neutrophil count > 1.5 x 109/L
   * Platelets >100 x 109/L
   * Serum creatinine ≤ 2.0 x ULN (upper limit of normal)
   * Serum bilirubin ≤ 1.5 x ULN
   * AST and ALT ≤ 2.5 x ULN (without liver metastasis), ≤ 5.0 x ULN (with liver metastasis)
8. Life expectancy ≥ 12 weeks at day 1

Exclusion Criteria:

1. Previous treatment with sunitinib or other VEGF-TKIs
2. Any major operation or irradiation within 4 weeks of baseline disease assessment
3. Any clinically significant gastrointestinal abnormalities which may impair intake or absorption of the study drug
4. CNS metastasis with continuous corticosteroid use within 4 weeks of baseline disease assessment (Asymptomatic CNS metastasis patients can be enrolled)
5. Patients with uncontrolled or significant cardiovascular disease (AMI within 12 months, Unstable angina within 6 months, NYHA Class III, IV Congestive heart failure or left ventricular ejection fraction below local institutional lower limit of normal or below 45%, Congenital long QT syndrome, Any significant ventricular arrhythmia, Any uncontrolled second or third degree heart block, Uncontrolled hypertension)
6. Concomitant malignancy (except adequately treated basal cell cancer of skin or cervical cancer in situ)
7. Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
8. Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into this trial. (including active bleeding, untreated DVT or thromboembolism)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Up to 6 months
  CR or PR by RECIST criteria version 1.1

SECONDARY OUTCOMES:
Disease control rate | Up to 6 months
  CR or PR or SD by RECIST criteria version 1.1
Progression-Free Survival | Up to 6 months
Overall survival | From first day of study treatment to day of any kind of death, assessed up to 24 months
Incidence of treatment related adverse events [Safety and Tolerability] | Up to 6 months
  Number of patients with adverse events during cycle 1 (each cycle is 21 days). Subjects will be evaluated for toxicity according to NCI-CTCAE(Common Terminology Criteria for Adverse Events) of version 4.0.

OTHER OUTCOMES:
Biomarker endpoint | Day 1
  When available, banked tumor tissue for genomic analysis for predictive biomarker of sunitinib.

CONTACTS AND LOCATIONS:
Overall Officials: Jong Seok Lee, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

REFERENCES:
- See also: Oral Presentation at WCLC 2018 (OA11.05 ) — https://doi.org/10.1016/j.jtho.2018.08.297